CLINICAL TRIAL: NCT04730570
Title: Essential Coaching for Every Mother: A Randomized Controlled Trial Evaluating an Text Message Postpartum Program for Mothers
Brief Title: Essential Coaching for Every Mother, a Postpartum Text Message Program for Canadian Mothers
Acronym: ECEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Justine Dol, Principal Investigator, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1024984
Record Dates: First submitted 2021-01-19; First posted 2021-01-29 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Maternal Distress
Keywords: maternal self-efficacy; postpartum depression; postpartum anxiety; mobile health education; postpartum support
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: The current study is a 2-group parallel arm randomized controlled trial, stratified by parity.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Blinding is not possible for participants and thus participants will be informed of their group allocation.
  To minimize personnel blinding related to data collection, no hospital staff (nurse midwives, physicians, other healthcare providers) are required to be aware of participant's involvement in the study. This is possible as Essential Coaching for Every Mother is sent to the participant's personal cell phone with no intervention occurring in person.
  The PI will be aware of participant allocation and will be responsible for collecting data but will not be involved in the randomization procedure which occurs directly in the TextIt platform. Additionally, there is no interaction with the participants from the PI or anyone on the research team as everything occurs remotely via a previously set up process, reducing any risk of influencing participant response and influencing outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential Coaching for Every Mother Intervention (Experimental): Women in the intervention arm will receive the Essential Coaching for Every Mother messages up to six-weeks postpartum. No changes in standard care.
  Interventions: Behavioral: Essential Coaching for Every Mother
- Standard care (No Intervention): Women in the control group will receive no content messages. No changes in standard care.

INTERVENTIONS:
Behavioral: Essential Coaching for Every Mother — Essential Coaching for Every Mother consists of 53 standardized text messages that provide evidence-based information that women should be aware of related to caring for their newborn and maternal mental health. Messages are personalized with the name of the child. Messages sent from birth to six-weeks postpartum, with two messages sent per day in the first two weeks and a daily message for weeks 3-6. The following topics covered in Essential Coaching for Every Mother include anxiety, depression, maternal self-care, postnatal follow-up, breastfeeding or formula feeding, infant concerns, cord care, well-baby care, normal development, crying, and safe sleep. Women who receive the messages will be able to self-select breastfeeding or formula feeding messages.
  Arms: Essential Coaching for Every Mother Intervention

SUMMARY:
The purpose of this study is to evaluate a text message-based program called Essential Coaching for Every Mother which sends daily text messages during the immediate six-week postnatal period. Essential Coaching for Every Mother consists of standardized text messages that provide evidence-based information that women should be aware of related to caring for their newborn and maternal mental health.

DETAILED DESCRIPTION:
This is a 2-group parallel arm randomized controlled trial. Participants will be randomized into either the intervention or a control group, stratified by parity. No changes to in-person care will occur.

Mothers in the intervention group will receive daily text messages from enrollment after birth until six-weeks postpartum.

Mothers in the control group will receive no content messages.

Mothers will be recruited both antenatally and postnatally through social media and study posters. All recruitment and participant engagement will occur remotely via text message. Women who are 37+ weeks pregnant up to 10 days postpartum will be eligible to send a text to a study specific number and complete an eligibility screening. If determined eligible once they deliver, the participant will be randomized into the intervention or control group and they will be asked to complete an electronic consent form and the baseline survey. Participants in the intervention group will start receiving the Essential Coaching for Every Mother program based on their delivery date up to six weeks postpartum. Mothers in the control group will only receive reminder texts to complete the follow-up surveys. Both groups will be asked to complete an online survey at enrolment, six-weeks and six-months postpartum.

The investigators aim to recruitment 140 participants in total, 70 per group.

ELIGIBILITY:
Inclusion Criteria:

To enroll antenatally, participants must:

* be at least 37 weeks pregnant
* have daily access to a mobile phone with text message capabilities
* are over 18 years of age
* speak and read English
* live in Nova Scotia, Canada.

To enroll postnatally, participants must:

* have an infant under 10 days of age
* have daily access to a mobile phone with text message capabilities
* are over 18 years of age
* speak and read English
* live in Nova Scotia, Canada.

Exclusion Criteria:

* newborn die or are expected to die prior to leaving the hospital
* they have no access to mobile phone, either personal or shared
* unwilling to receive text messages
* decline or withdraw to participate
* participated in Phase I of this project.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Self Efficacy | Change from enrolment (baseline) to six-weeks
  Karitane Parenting Confidence Scale (Minimum: 0, Maximum: 45; Higher score indicates greater self-efficacy)

SECONDARY OUTCOMES:
Social support | Change from enrolment (baseline) to six-weeks
  Multidimensional Scale of Perceived Social Support (For the sub-scales of family, friends, and significant other [Minimum: 0, Maximum: 4]; for the total score, [Minimum: 0, Maximum: 12]; higher scores indicate greater support).
Postpartum anxiety | Change from enrolment (baseline) to six-weeks
  Postpartum Specific Anxiety Scale (Minimum: 51, Maximum: 204; Higher score indicates higher anxiety)
Postpartum depression | Change from enrolment (baseline) to six-weeks
  Edinburgh Postnatal Depression Scale (Minimum: 0, Maximum: 30; Higher score indicates higher depression)
Self-Efficacy | Change from six-weeks to six-months postpartum
  Karitane Parenting Confidence Scale (Minimum: 0, Maximum: 45; Higher score indicates greater self-efficacy)
Social Support | Change from six-weeks to six-months postpartum
  Multidimensional Scale of Perceived Social Support (For the sub-scales of family, friends, and significant other [Minimum: 0, Maximum: 4]; for the total score, [Minimum: 0, Maximum: 12]; higher scores indicate greater support).
Postpartum anxiety | Change from six-weeks to six-months postpartum
  Postpartum Specific Anxiety Scale (Minimum: 51, Maximum: 204; Higher score indicates higher anxiety)
Postpartum depression | Change from six-weeks to six-months postpartum
  Edinburgh Postnatal Depression Scale (Minimum: 0, Maximum: 30; Higher score indicates higher depression)

OTHER OUTCOMES:
Implementation extent (Reach) | Through study completion, an average of 1 year
  What was the reach (i.e., enrolment rate)?
Implementation extent (completion) | Through study completion, an average of 6 weeks
  What was the completion rate (e.g., withdrawal rate)?
Implementation extent (dose) | Through study completion, an average of 6 weeks
  What was the dose received (i.e., number of messages received)?
Implementation quality | 6-weeks postpartum
  Qualitative feedback on program:
  * What did you like most about Essential Coaching for Every Mother? [open ended]
  * What did you like least about Essential Coaching for Every Mother? [open ended]
  * Did you face any barriers with acting on the information received from Essential Coaching for Every Mother at home (e.g., geographical impacts, cellular access, health seeking opportunities)? If yes, please describe. [open ended]
  * How can Essential Coaching for Every Mother be improved further? [open ended]

CONTACTS AND LOCATIONS:
Overall Officials: Justine Dol, MSc, Principal Investigator — Dalhousie University
Locations (1):
- IWK Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dol J, Aston M, McMillan D, Tomblin Murphy G, Campbell-Yeo M. Effectiveness of a Postpartum Text Message Program (Essential Coaching for Every Mother) on Maternal Psychosocial Outcomes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Mar 25;10(3):e27138. doi: 10.2196/27138. PMID 33764309
- [Background] Dol J, Aston M, McMillan D, Tomblin Murphy G, Campbell-Yeo M. Participants' Perceptions of Essential Coaching for Every Mother-a Canadian Text Message-Based Postpartum Program: Process Evaluation of a Randomized Controlled Trial. JMIR Form Res. 2022 May 13;6(5):e36821. doi: 10.2196/36821. PMID 35559855
- [Result] Dol J, Tomblin Murphy G, Aston M, McMillan D, Campbell-Yeo M. Design, development and usability testing of Essential Coaching for Every Mother: A postnatal text message educational intervention. Women Birth. 2021 May;34(3):e228-e236. doi: 10.1016/j.wombi.2020.05.004. Epub 2020 May 29. PMID 32475782